CLINICAL TRIAL: NCT04385771
Title: Cytokine Adsorption in Patients With Severe COVID-19 Pneumonia Requiring Extracorporeal Membrane Oxygenation - Randomized, Controlled, Open-label Intervention, Multi-center Trial (CYCOV-II-study)
Brief Title: Cytokine Adsorption in Patients With Severe COVID-19 Pneumonia Requiring Extracorporeal Membrane Oxygenation
Acronym: CYCOV-II
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: security concerns based on preliminary results from preceding CYCOV-I-study suggesting higer mortality in cytokine adsorption group
Sponsor: Dr. Alexander Supady (Other)
Collaborators: Klinikum Ibbenbüren (Unknown); Ludwig-Maximilians - University of Munich (Other); University Hospital, Saarland (Other); Klinikum Ludwigsburg (Other); University of Ulm (Other); SLK Kliniken Heilbronn GmbH (Other); Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Sponsor-Investigator, Dr. Alexander Supady, Attending Physician - Oberarzt, University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYCOV-II
Record Dates: First submitted 2020-04-19; First posted 2020-05-13 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus Infection; COVID; SARS-CoV 2; Respiratory Failure; Cytokine Storm; Extracorporeal Membrane Oxygenation
Keywords: COVID-19; ECMO; ARDS; Cytokine Adsorption
MeSH Terms: conditions — Coronavirus Infections; Respiratory Insufficiency; Cytokine Release Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: randomized controlled trial examining COVID-patients requiring vv-ECMO therapy (+/- cytokine adsorption)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vv-ECMO + cytokine adsorption (Experimental): after indication of treatment with vv-ECMO in acute respiratory failure in COVID-19-disease, patients will additionally receive cytokine adsorption using a Cytosorb adsorber
  Interventions: Device: vv-ECMO + cytokine adsorption (Cytosorb adsorber)
- vv-ECMO (no cytokine adsorption) (Other): treatment with vv-ECMO in acute respiratory failure in COVID-19-disease (standard treatment without additional cytokine adsorption)
  Interventions: Device: vv-ECMO only (no cytokine adsorption)

INTERVENTIONS:
Device: vv-ECMO + cytokine adsorption (Cytosorb adsorber) — in COVID-19-diseased vv-ECMO patients additional treatment with cytokine adsorption using a Cytosorb adsorber will be randomized (vs. control group)
  Arms: vv-ECMO + cytokine adsorption
Device: vv-ECMO only (no cytokine adsorption) — COVID-19-diseased treated with vv-ECMO
  Arms: vv-ECMO (no cytokine adsorption)

SUMMARY:
In December 2019 in the city of Wuhan in China, a series of patients with unclear pneumonia was noticed, some of whom have died of it. In virological analyses of samples from the patients' deep respiratory tract, a novel coronavirus was isolated (SARS-CoV-2). The disease spread rapidly in the city of Wuhan at the beginning of 2020 and soon beyond in China and, in the coming weeks, around the world.

Initial studies described numerous severe courses, particularly those associated with increased patient age and previous cardiovascular, metabolic and respiratory diseases. A small number of the particularly severely ill patients required not only highly invasive ventilation therapy but also extracorporeal membrane oxygenation (vv-ECMO) to supply the patient's blood with sufficient oxygen.

Even under maximum intensive care treatment, a very high mortality rate of approximately 80-100% was observed in this patient group. In addition, high levels of interleukin-6 (IL-6) could be detected in the blood of these severely ill patients, which in turn were associated with poor outcome.

From experience in the therapy of severely ill patients with severe infections and respiratory failure, we know that treatment with a CytoSorb® adsorber can lead to a reduction of the circulating pro- and anti-inflammatory cytokines and thus improve the course of the disease and the outcome of the patients.

The aim of the study is to investigate the influence of extracorporeal cytokine adsorption on interleukin-6-levels and time to successful ECMO explantation under controlled conditions in patients with particularly severe COVID-19 disease requiring extracorporeal membrane oxygenation.

DETAILED DESCRIPTION:
In December 2019, a series of unexplained cases of pneumonia in the city of Wuhan in China has come to light. In virologic analyses of samples from the patients' deep respiratory tract, a novel coronavirus was isolated (first named 2019-nCoV, then SARS-CoV-2). The disease spread rapidly in the city of Wuhan in early 2020 and soon beyond. On 30 January 2020, the Director-General of the World Health Organization (WHO) declared the outbreak a public health emergency of international concern, and on 11 March 2020, the World Health Organization declared the virus a pandemic.

In humans, an infection with the virus can cause respiratory tract infections or even very severe pneumonia - these often end fatally, especially in old and pre-diseased patients. Due to the novelty of the virus, the data basis for therapy is very limited. To date, there are no clinical data for an effective specific therapy, nor is there a vaccination against the virus available, so that therapy, especially intensive care treatment for very severe courses, must concentrate only on supportive treatment of lung failure and other complications.

The virus is highly contagious and infection results in a relevant number of deaths. Due to very uncertain data on the spread of the virus in the population, it is difficult to estimate the mortality rate - the case fatality rate is about 4% based on the known case numbers.

In reports on the treatment of the first cases in Wuhan (Hubei Province, China) in January 2020, the need for intensive care treatment is described for about a quarter of the inpatient cases, 10-17% had to be ventilated invasively, and veno-venous extracorporeal membrane oxygenation (vv-ECMO) was necessary in 2-4% of the inpatient cases. Patients requiring ECMO have an extremely high mortality rate of 83-100% in the studies published, so far.

In severe cases a pronounced release of vasoactive cytokines was repeatedly observed. Excessive release of these vasoactive mediators ("cytokine storm") can result in severe vasodilatation and membrane leakage, which can ultimately lead to vasoplegic shock that is difficult to control. Ruan et al. and Zhou et al. have identified high interleukin 6 (IL-6) levels as a potential predictor of a fatal outcome when compared between survivors and patients who died of COVID-19 disease.

IL-6 is also an important factor in the pathophysiology of severe septic shock and excessive immune response in hemophagocytic lymphohistiocytosis (HLH) - for both indications has been shown, that the extracorporeal adsorption of IL-6 and other vasoactive substances in a CytoSorb® adsorber (CytoSorbents Corporation, Monmouth Junction, NJ, USA) leads to a significant reduction of these cytokines in the patient blood. Clinical experience and (previously unpublished) data from our monocentric registry study show that cytokine adsorption in a CytoSorb® Adsorber can also be safely integrated into a vv-ECMO system.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2-infection with COVID-pneumonia
* vv-ECMO therapy

Exclusion Criteria:

* known patient will against participation in the study or against the measures applied in the study
* a decision (made prior to inclusion of the patient into this trial) to terminate the treatment within the next 24 hours

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
IL-6 reduction by 75% or more after 72 hours as compared to the baseline measurement | 72 hours
  measurement of IL-6 levels in patient blood after 72 hours of cytokine adsorption (in relation to level before initiation of cytokine adsorption)
time to successful ECMO-explantation | 30 days
  time to successful ECMO-explantation within 30 days after randomization

SECONDARY OUTCOMES:
Ventilator free days (VFD) | 30 days
  Ventilator free days (VFD) in the first 30 days after randomization, where invasive mechanical ventilation (IMV), non-invasive ventilation (NIV) and ECMO are defined as ventilator days. VFD=0, if the patient dies in the first 30 days after randomization
Time to extubation from ventilation and explantation from ECMO | 30 days
  Time to extubation from ventilation and explantation from ECMO. Death under ventilation and/or ECMO will be analyzed as a competing event. The time will be censored at the time of last visit for surviving patients under ventilation and/or ECMO.
Overall survival time | 30 days
  Overall survival time, defined as time from randomization to death. The time will be censored at the time of last visit for surviving patients.
Days on intensive care unit (ICU) | 30 days
  Days on intensive care unit (ICU)
Vasopressor dosage | 24, 48, 72 hours
  Vasopressor dosage of adrenaline, noradrenaline, vasopressin, and dobutamine at 24, 48,72 h
Fluid substitution and fluid balance | 24, 48, 72 hours
  Total fluid[ml] substitution and fluid balance [ml] at 24, 48, 72 h
Serum lactate | 24, 48, 72 hours
  Serum lactate at 24, 48, 72 h
Urine output | 24, 48, 72 hours
  Urine output at 24, 48, 72 h
Willebrand factor | 24, 48, 72 hours
  Willebrand factor at 24, 48, 72 h
d-dimers | 24, 48, 72 hours
  d-dimers at 24, 48, 72 h
interleukin-6 levels | 24, 48, 72 hours
  interleukin-6 levels at 24, 48, 72 h
SOFA-Score | 24, 48, 72 hours
  Sequential Organ Failure Assessment Score at 24, 48, 72 h (values from 6 to 24, where the higher values explain higher disease severity)
serious adverse device effects | 30 days
  serious complications or malfunctions related to the CytoSorb device
adverse event of special interest: air in the ECMO system | 30 days
  unintended air in the ECMO system during operation of the device
adverse event of special interest: blood-clotting in the ECMO system | 30 days
  unintended blood-clotting in the ECMO system during operation of the device
adverse event of special interest: bleeding complications | 30 days
  major bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Supady, Dr., MPH, Principal Investigator — University Clinic Freiburg
Locations (3):
- Germany (3):
  - University Clinic Freiburg, Freiburg im Breisgau
  - Klinikum Ibbenbueren, Ibbenbueren
  - Klinikum Ludwigsburg, Ludwigsburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shekar K, McAuley DF, Brodie D. Cytokine adsorption during ECMO for COVID-19-related ARDS. Lancet Respir Med. 2021 Jul;9(7):680-682. doi: 10.1016/S2213-2600(21)00207-1. Epub 2021 May 14. No abstract available. PMID 34000235
- [Derived] Rieder M, Duerschmied D, Zahn T, Lang C, Benk C, Lother A, Biever P, Bode C, Wengenmayer T, Staudacher D, Supady A. Cytokine Adsorption in Severe Acute Respiratory Failure Requiring Veno-Venous Extracorporeal Membrane Oxygenation. ASAIO J. 2021 Mar 1;67(3):332-338. doi: 10.1097/MAT.0000000000001302. PMID 33627609
- [Derived] Rieder M, Schubach F, Schmoor C, von Spee-Mayer C, Wengenmayer T, Rilinger J, Staudacher D, Bode C, Duerschmied D, Supady A. Cytokine adsorption in patients with severe COVID-19 pneumonia requiring extracorporeal membrane oxygenation: protocol for a randomised, controlled, open-label intervention, multicentre trial. BMJ Open. 2021 Jan 17;11(1):e043345. doi: 10.1136/bmjopen-2020-043345. PMID 33455938